CLINICAL TRIAL: NCT05391126
Title: GENOCARE: A Prospective, Randomized Clinical Trial of Genotype-Guided Dosing Versus Usual Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reema A. Patel (Other)
Responsible Party: Sponsor-Investigator, Reema A. Patel, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MCC-22-GI-125-PMC
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Pancreatic Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genocare Guided (Experimental)
  Interventions: Drug: Irinotecan
- Usual Care (No Intervention)

INTERVENTIONS:
Drug: Irinotecan — Usual dosing per package insert.
  Other Names: Nano-liposomal Irinotecan; Onyvide
  Arms: Genocare Guided

SUMMARY:
This is a prospective, randomized study designed to compare genotype-guided dosing to usual care in patients with pancreas cancer and colorectal cancer who are UGT1A1 intermediate metabolizers (*1/*28) (heterozygotes) and usual UGT metabolizers (*1/*1). All patients will be assessed for UGT1A1 genotype at screening and those with intermediate or usual UGT1A1 genotypes (*1/*28, *1/*1) will be randomized to genotype-guided dosing versus usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed stage I-IV pancreas or stage III-IV colorectal cancer who are planning to undergo treatment.
* Prior treatment is allowed, specifically surgery and/or radiation and non-irinotecan containing regimens are allowed.
* Age ≥ 18 years.
* ECOG performance status ≤ 1.
* Patients must have adequate organ and marrow function as defined below:
* Measurable or non-measurable disease.

Exclusion Criteria:

* Patients who received prior treatment with irinotecan are excluded.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with targeted therapy, in the opinion of the treating physician.
* Pregnant women are excluded from this study.
* Patients who are not planned for treatment of their cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Events Frequency | 6 months
  To compare the frequency of cycle 1 grade 3-5 adverse effects in individuals with a *1/*28 or *1/*1 genotype who receive genotype-guided dosing and to those who are randomized to receive usual care.

SECONDARY OUTCOMES:
Overall Survival | 5 years
  To evaluate overall survival between individuals randomized to receive genotype-guided dosing and those who are randomized to receive usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Reema A Patel, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No